CLINICAL TRIAL: NCT03182647
Title: Long-term Follow-up of Anterior Cruciate Ligament Injury
Acronym: ACLLTFU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Joanna Kvist, Professor, Linkoeping University
Other Study IDs: ACL LTFU
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non surgery: Patients were not treated with surgery initially
  Interventions: Other: Non surgical initial ACL treatment
- Surgery: Patients had an initial surgical treatment
  Interventions: Procedure: Surgically treatment of the ACL

INTERVENTIONS:
Procedure: Surgically treatment of the ACL — Surgical initial ACL treatment
  Groups: Surgery
Other: Non surgical initial ACL treatment — Non surgical initial ACL treatment
  Groups: Non surgery

SUMMARY:
Anterior cruciate ligament (ACL) rupture is one of the most common sports-related knee injuries. Because it is such a significant injury - requiring a long period of rehabilitation before the injured person is ready to return to physical activity, the burden of injury is high. This can help to explain why so much of orthopaedic research is devoted to evaluating the outcomes of ACL injury. However, while there has been extensive study of short-term (up to 5 years after injury) outcomes, few studies have followed patients beyond 15 years after their ACL injury. This is important because long-term follow-up can provide key insights to guide the information provided to newly injured patients (e.g. to help set realistic expectations of what the injured person can expect of their knee function in the future), and help us evaluate the efficacy of previous treatments.

The primary aim is to assess the influence of an acute ACL injury on knee function and quality of life, 32-37 years after the index injury. Approximately 300 patients injured between 1980 and 1985 will be invited to participate in the study. Patient- and clinician-reported outcomes, and radiographic osteoarthritis will be evaluated.

DETAILED DESCRIPTION:
Patients injuring their ACL between 1980 and 1985 have periodically been followed since the injury. Now, we plan to contact all patients and invite them to participate. The patients will be asked to

1. complete a questionnaire battery
2. visit the movement laboratory at Linköping University for an objective assessment of knee function and
3. have an x-ray of both knee joints.

Baseline information including associated injuries, treatment and activity level exist for all the patients. At that time, rehabilitation was normally completed after 4-6 months for non-operatively treated patients, and nine months after ACL surgery.

ELIGIBILITY:
Inclusion Criteria:

* primary ACL injury between 1980 and 1985, age between 15 and 40 at injury

Exclusion Criteria:

* all patients from the initial cohort will be invited for participation

Ages: 47 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Baseline data from the time for injury were collected consequently. The initial 167 patients were included in a randomised clinical trial of surgical vs. non-surgical treatment and the following patients were treated according to common practise at that time.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Self reported knee function | 32-37 years after ACL injury
  Knee Injury and Osteoarthritis Outcome Score, KOOS 4 (Pain, Symptoms, Sport/Rec, QOL subscales)
Osteoarthritis | 32-37 years after ACL injury
  Development of osteoarthritis examined with tibiofemoral and patellofemoral radiographs

SECONDARY OUTCOMES:
Quality of life | 32-37 years after ACL injury
  ACL-Quality of Life scale (ACL-QoL)
Physical activity | 32-37 years after ACL injury
  Total time over the previous week spent doing moderate, and vigorous activity AND accelerometer measures
Objective assessment of knee function | 32-37 years after ACL injury
  Concentric isokinetic muscle strength
Objective assessment of knee function | 32-37 years after ACL injury
  Functional testing; stand-up test
Objective assessment of knee function | 32-37 years after ACL injury
  Functional testing; hopping performance in one leg hop for distance
Objective assessment of knee function | 32-37 years after ACL injury
  Postural control (one leg stand test)
Associated injuries and additional surgery | 32-37 years after ACL injury
  Patient reported

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kvist, Professor, Principal Investigator — IMH Linkoping University, Sweden
Locations (1):
- Linkoping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meunier A, Odensten M, Good L. Long-term results after primary repair or non-surgical treatment of anterior cruciate ligament rupture: a randomized study with a 15-year follow-up. Scand J Med Sci Sports. 2007 Jun;17(3):230-7. doi: 10.1111/j.1600-0838.2006.00547.x. PMID 17501866
- [Result] Andersson C, Odensten M, Gillquist J. Knee function after surgical or nonsurgical treatment of acute rupture of the anterior cruciate ligament: a randomized study with a long-term follow-up period. Clin Orthop Relat Res. 1991 Mar;(264):255-63. PMID 1997243
- [Derived] Filbay S, Andersson C, Gauffin H, Kvist J. Prognostic Factors for Patient-Reported Outcomes at 32 to 37 Years After Surgical or Nonsurgical Management of Anterior Cruciate Ligament Injury. Orthop J Sports Med. 2021 Aug 11;9(8):23259671211021592. doi: 10.1177/23259671211021592. eCollection 2021 Aug. PMID 34395684
- [Derived] Kvist J, Filbay S, Andersson C, Ardern CL, Gauffin H. Radiographic and Symptomatic Knee Osteoarthritis 32 to 37 Years After Acute Anterior Cruciate Ligament Rupture. Am J Sports Med. 2020 Aug;48(10):2387-2394. doi: 10.1177/0363546520939897. PMID 32736511